CLINICAL TRIAL: NCT04818905
Title: Effects of Helichrysum Italicum Infusion on Resting Energy Expenditure and Fat Oxidation in Humans
Brief Title: Helichrysum Italicum Infusion Ingestion in Humans
Acronym: SMILJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Responsible Party: Principal Investigator, Zala Jenko Praznikar, Associate professor, University of Primorska
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SMILJ_pilot
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Energy Expenditure; Substrate Oxidation; Blood Pressure
Keywords: bioactive compounds; functional beverages; metabolism; helath

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Helichrysum italicum infusion (Experimental): 1 g of milled plant material (Helichrysum italicun) immersed in hot water (200 mL, 100 °C) for 10 minutes.
  Interventions: Dietary Supplement: Helichrysum italicum infusion
- Hot water (Placebo Comparator): The control beverage contained only hot water (200 mL, 100 ˚C).
  Interventions: Other: Hot water

INTERVENTIONS:
Dietary Supplement: Helichrysum italicum infusion — Active beverage or control beverage consumption after overnight fasting and calorimetry measurement on a single subject. After seven days washout period follows the consumption of the alternate beverage and measurements.
  Other Names: Active beverage
  Arms: Helichrysum italicum infusion
Other: Hot water — Active beverage or control beverage consumption after overnight fasting and calorimetry measurement on a single subject. After seven days washout period follows the consumption of the alternate beverage and measurements.
  Other Names: Control beverage
  Arms: Hot water

SUMMARY:
The study evaluates the acute effects of Helichrysum italicum on resting energy expenditure and substrate oxidation in humans. The resting energy expenditure and substrate oxidation will be measured by indirect calorimetry at baseline and after ingestion of either Helichrysum italicum infusion or hot water.

DETAILED DESCRIPTION:
Bioactive compounds found in medicinal plants and plant extracts, such as polyphenols, represent the oldest and most widely used form of alternative or complementary treatments for the prevention and management of obesity. Their consumption is currently increasing in the population due to the high cost, potential adverse effects and limited benefits of currently available pharmaceutical drugs. Helichrysum italicum is a mediterranean plant with promising nutraceutical activities. The plant is known as a rich source of biologically active compounds such as polyphenolic antioxidants, which are recognized in the prevention of various non-communicable chronic diseases. However, most of its traditionally claimed uses have not yet been scientifically proven.

The proposed study will investigate the acute effect of Helichrysum italicum infusion on resting energy expenditure, substrate oxidation, respiratory quotient and blood pressure in a pilot study of 11 male adults. It will be designed as a crossover study. Half of the participants will consume the Helichrysum italicum infusion and the other half will consume hot water. After seven days of washout period the participants will consume the alternate beverage.

ELIGIBILITY:
Inclusion Criteria:

* healthy, weight-stable (±3 kg in the last 3 months), normotensive, non-smokers, no use of dietary supplements or frequent use of medication and no known metabolic disorders.

Exclusion Criteria:

* females, smoking, medications, dietary supplements, metabolic diseases, hypertensive

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 11 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in resting energy expenditure | Change from baseline to 30 minutes and 120 minutes.
  Resting energy expenditure will be determined with indirect calorimetry.
Changes in fat oxidation | Change from baseline to 30 minutes and 120 minutes.
  Substrate oxidation will be determined with indirect calorimetry.
Respiratory quotient | Change from baseline to 30 minutes and 120 minutes.
  Respiratory quotient will be determined with indirect calorimetry.
Blood pressure | Change from baseline to 30 minutes and 120 minutes.
  Systolic and diastolic blood pressures will be determined with blood pressure device (Omron M3)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Primorska, Faculty of Health Sciences, Izola, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Konstantinidi M, Koutelidakis AE. Functional Foods and Bioactive Compounds: A Review of Its Possible Role on Weight Management and Obesity's Metabolic Consequences. Medicines (Basel). 2019 Sep 9;6(3):94. doi: 10.3390/medicines6030094. PMID 31505825
- [Background] Manach C, Scalbert A, Morand C, Remesy C, Jimenez L. Polyphenols: food sources and bioavailability. Am J Clin Nutr. 2004 May;79(5):727-47. doi: 10.1093/ajcn/79.5.727. PMID 15113710
- [Background] Antunes Viegas D, Palmeira-de-Oliveira A, Salgueiro L, Martinez-de-Oliveira J, Palmeira-de-Oliveira R. Helichrysum italicum: from traditional use to scientific data. J Ethnopharmacol. 2014;151(1):54-65. doi: 10.1016/j.jep.2013.11.005. Epub 2013 Nov 14. PMID 24239849
- [Background] Soga S, Ota N, Shimotoyodome A. Stimulation of postprandial fat utilization in healthy humans by daily consumption of chlorogenic acids. Biosci Biotechnol Biochem. 2013;77(8):1633-6. doi: 10.1271/bbb.130147. Epub 2013 Aug 7. PMID 23924724
- [Derived] Kenig S, Kramberger K, Petelin A, Bandelj D, Baruca Arbeiter A, Miklavcic Visnjevec A, Peeters K, Mohorko N, Sik Novak K, Jenko Praznikar Z. Helichrysum italicum ssp. italicum Infusion Promotes Fat Oxidation in Hepatocytes and Stimulates Energy Expenditure and Fat Oxidation after Acute Ingestion in Humans: A Pilot Study. Plants (Basel). 2021 Jul 23;10(8):1516. doi: 10.3390/plants10081516. PMID 34451560